CLINICAL TRIAL: NCT04548505
Title: Recovery of Exertion Ability Following COVID-19 Infection in Military Staff
Acronym: CovEx
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-30; 2020-A02140-39 (Other: IDRCB)
Record Dates: First submitted 2020-09-11; First posted 2020-09-14 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV Infection
Keywords: physical activity
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Paris Fire Brigade staff have been particularly exposed to COVID-19 due to rescue and care activities for victims at risk in Paris area (where the virus was actively circulating). In addition, when the pandemic began in France, they had to take care of patients before procedures to protect caregivers were implemented.

The contamination of young military personnel, whose physical capacity was put into strain at work, raises the question of the consequences of COVID-19 on their physical fitness. At the time, the medium- and long-term evolution of this disease and its possible repercussions on physical fitness are unknown. Moreover, like any soldiers who have been confined, they may present at least a cardio-respiratory deconditioning (sometimes independent of the disease making it difficult to distinguish between a sequelae of the infection or rehabilitation).

Based on previous coronavirus epidemics (Sars-Cov 1 and Mers-Cov), it appears that long-term sequelae are possible even in mild forms and can result in an alteration of exertion ability.

In the current context and in the absence of national or international recommendations on the return to physical activity, the French Armed Forces Health Service has proposed a simple management plan aiming at: i) allowing mass screening for possible exercise intolerance and targeting at-risk personnel, ii) allowing individualized re-training and iii) guaranteeing that military personnel can carry out their mission without jeopardizing their health.

ELIGIBILITY:
Inclusion Criteria:

* Be an active military personnel of the Paris Fire Brigade
* Be at least 18 years of age
* Benefiting or having benefited from the post-COVID medical care provided by the French Armed Forces Health Service

Exclusion Criteria:

* Be under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population is composed of active military personnel of the Paris Fire Brigade who have been infected with COVID-19 and thus are benefiting or have benefited from the post-COVID medical car provided bay the French Armed Forces Health Service.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-04-05 (Estimated); Study Completion 2023-04-05 (Estimated)

PRIMARY OUTCOMES:
Magnitude of the decrease in aerobic performance on return to work | Up to 18 months
  Aerobic performance will be assessed through a test called VAMEVAL. VAMEVAL consists of running around a track marked out every 50 meters to the rhythm of a soundtrack that accelerates at a rate of 0.5 km/h in 2-minute increments until exhaustion or inability to maintain the pace of the race. The result of the test made on return to work will be compared to the last result on the same test performed before COVID-19 infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided